CLINICAL TRIAL: NCT06752954
Title: Comparison of the Effectiveness of Viabahn® Vs. Drug-Coated Balloon With/without Bail-Out Bare Metal Stent in Treating Complicated Femoropopliteal Lesions
Brief Title: The Effectiveness of Covered Stent Viabahn and Drug-coated Balloon for Complex Femoropopliteal Artery Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, Chengzhi Li, Doctor of Medicine, First Affiliated Hospital of Jinan University
Other Study IDs: The support study
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Viabahn endoprosthesis; Drug-coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Viabahn endoprosthesis group: Patients underwent endovascular treatment for femoropopliteal lesions. The lesion will be treated by Viabahn endoprosthesis.
  Interventions: Device: Viabahn endoprosthesis group
- Drug-coated balloon group: Patients underwent endovascular treatment for femoropopliteal lesions. The lesion will be treated by drug-coated balloon.
  Interventions: Device: Drug-coated balloon group

INTERVENTIONS:
Device: Viabahn endoprosthesis group — Viabahn endoprosthesis group：Patients underwent endovascular treatment for femoropopliteal lesions. The lesion will be treated by Viabahn endoprosthesis.
  Groups: Viabahn endoprosthesis group
Device: Drug-coated balloon group — Patients underwent endovascular treatment for femoropopliteal lesions. The lesion will be treated by drug-coated balloon.
  Groups: Drug-coated balloon group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the covered stent Viabahn in treating long de novo femoropopliteal lesions (stenosis ≥ 25 cm, total occlusion ≥ 15 cm) or in-stent restenosis compared to drug-coated balloons (DCB) with or without a bailout bare nitinol stent.

DETAILED DESCRIPTION:
This is a multicenter, observational prospective cohort clinical trial with clinical and image follow-up for two years post-procedure. Approximately 200 subjects will be enrolled into a Viabahn group (observe arm) or drug-coated balloons (DCB) group (contrast arm); Each group will include 100 patients.

All enrolled patients will be followed up for 12 and 24 months to assess the incidence of restenosis by duplex ultrasound and major adverse events. Follow-up visits occur at 12 and 24 months, as well as telephone visits after 1, 3,6 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥ 18 years old.
2. Patient understands the nature of the procedure and provides written informed consent before enrolment in the study
3. The patient is willing to comply with specified follow-up evaluations at the specified times.
4. The patient presented a score from 2 to 5 following Rutherford classification.
5. The patient has a projected life expectancy of at least 24 months
6. Subject has a de novo or restenotic lesion with ≥ 70% stenosis in femoropopliteal artery, and for de novo lesion, the total lesion length ≥ 25cm, or chronic total occlusion (CTO) length ≥15cm.

Exclusion Criteria:

1. Patients with known hypersensitivity or contraindication to any of the following medications: Contrast media, Nitinol-titanium, antiplatelet therapy, anticoagulants, or thrombolytics therapy
2. Pregnant women or Female patients with potential childbearing
3. Patients who exhibit acute intraluminal thrombus at the target lesion vessel
4. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
5. The patient is currently participating in another investigational drug or device study that interferes with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The patient is ≥ 18 years old.
  2. Patient understands the nature of the procedure and provides written informed consent before enrolment in the study
  3. The patient is willing to comply with specified follow-up evaluations at the specified times.
  4. The patient presented a score from 2 to 5 following Rutherford classification.
  5. The patient has a projected life expectancy of at least 24 months
  6. Subject has a de novo or restenotic lesion with ≥ 70% stenosis in femoropopliteal artery, and for de novo lesion, the total lesion length ≥ 25cm, or chronic total occlusion (CTO) length ≥15cm.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12-month
  Peak systolic velocity ratio (PSVR ≤2.4) without any repeat intervention.
Freedom from a composite of Major adverse events (MAEs) | 12-month
  Freedom from MAEs is defined as freedom from clinically-driven target vessel revascularization (CD-TVR), major amputation, and all-cause of death

SECONDARY OUTCOMES:
Procedural success | Immediately after interventional surgery
  Procedural success is defined as technical or device success without major adverse events during the hospital stay.
Primary assisted patency | 12-month
  Primary assisted patency is defined as maintaining patency in the target vessel after a repeat intervention to regain patency prior to complete occlusion.
Secondary patency | 12-month
  Secondary patency is defined as maintaining patency in the target vessel after a repeat intervention to correct complete occlusion in the treated arterial segment.
Clinically-driven target vessel revascularization (CD-TVR) | 12-month
  clinically-driven target vessel revascularization (CD-TVR) is defined as repeat intervention performed during enrollment in the clinical study.
Primary sustained clinical improvement | 12-month
  Defined as a sustained upward shift of at least one category on the Rutherford classification without the need for repeated target lesion revascularization (TLR) in surviving patients.
Secondary sustained clinical improvement | 12-month
  Defined as a sustained upward shift of at least one category on the Rutherford classification3, including the need for repeated target lesion revascularization (TLR) in surviving patients.
Vasc quality of life score | 12-month
  Change of Vasc quality of life score